CLINICAL TRIAL: NCT06895200
Title: CVS-Notifier - Smart Intraoperative Reminder to Implement Safety Principles in Laparoscopic Cholecystectomy
Brief Title: Smart Intraoperative Reminder to Implement Safety Principles in Laparoscopic Cholecystectomy
Acronym: CVS-Notifier
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IHU Strasbourg (Other)
Collaborators: Scialytics SAS (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 24-001
Record Dates: First submitted 2025-03-17; First posted 2025-03-26 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Cholecystectomy, Laparoscopic
Keywords: Laparoscopic cholecystectomy; Gallbladder; Safety; Critical View of Safety; CVS; Bile Duct Injuries; BDI

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study (Experimental)
  Interventions: Device: CVS-Notifier SaMD

INTERVENTIONS:
Device: CVS-Notifier SaMD — The CVS-Notifier SaMD reminds surgeons to time-out to check the CVS before the division of the cystic duct.

SUMMARY:
The Critical View of Safety (CVS) is universally recommended to prevent bile duct injuries in laparoscopic cholecystectomy. However, CVS is underutilized and bile duct injuries are not decreasing. The CVS-Notifier SaMD (Software as a Medical Device) reminds surgeons to verify the CVS before dividing the cystic duct, as recommended by guidelines. It is hypothesized that this systematic and timely reminder could improve the implementation of CVS without disturbing surgical workflows.

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy is the gold standard approach for the surgical removal of the gallbladder. However, between 0.3 and 1.5% of patients undergoing laparoscopic cholecystectomy experience a bile duct injury (BDI). This major complication translates into a threefold increase in mortality at 1 year, frequent medico-legal litigations, and an annual cost of about 1 billion dollars in the USA alone.

The visual perceptual illusion causing major BDIs can be prevented by implementing the Critical View of Safety (CVS). CVS consists of the clearance of the hepatocystic triangle from fat and connective tissue, the division of the lower part of the gallbladder from its liver bed, and ensuring that only two tubular structures-the cystic duct and the cystic artery-connected to the gallbladder are visible. Unfortunately, CVS implementation in surgical practices is as low as 9% and, in turn, BDIs do not decrease.

To improve the implementation of the CVS, multi-society consensus guidelines recommend to time-out to confirm CVS achievement before dividing cystic structures. A large quality improvement study demonstrated that a short time-out to recall CVS principles significantly increases CVS implementation rates. However, the implementation of the time-out and CVS decreases over time.

The CVS-Notifier SaMD reminds surgeons to time-out to verify the CVS before the division of the cystic duct. Such a systematic intraoperative reminder to implement best practices could help consistently perform safe laparoscopic cholecystectomies.

This first-in-human, exploratory study aims at evaluating the safety, usability, and potential impact of the CVS-Notifier SaMD in laparoscopic cholecystectomy.

The study is a single center, non-comparative, case series. Patients undergoing elective laparoscopic cholecystectomy who meet the eligibility criteria and express their consent to participate in the study will be enrolled. The CVS-Notifier SaMD will be installed on a medical grade computer connected to a secondary output of the laparoscopic video system (input) and to an auxiliary screen in the operating room (OR) (output). Surgeons will start the procedure as usual while the CVS-Notifier SaMD unobtrusively analyses the surgical video. When the beginning of the hepatocystic triangle dissection is detected, a visual reminder to verify CVS in an intraoperative time-out notification will appear on the auxiliary OR screen.

Surgeons and patients will be asked to fill in a survey to report their experience, after the procedure and before discharge, respectively.

Clinical, surgical, and device-related data will be collected and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman over 18 years old.
* Patient presenting with benign gallbladder disease requiring an elective laparoscopic cholecystectomy.
* Patient without contraindications to anaesthesia or laparoscopic cholecystectomy surgery.
* Patients capable of understanding and providing their written consent to the study.
* Patient affiliated to the French social security system.

Exclusion Criteria:

* Patients presenting with malignant gallbladder disease requiring an elective laparoscopic cholecystectomy.
* Pregnant or lactating patient.
* Patient in exclusion period (determined by a previous or a current study).
* Patient under guardianship or trusteeship.
* Patient under the protection of justice or deprived of liberty.
* Patient in situation of emergency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-03 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Rate of CVS-Notifier SaMD related complications | From the day of the procedure up to 30 days after surgery
  The rate of CVS-Notifier SaMD related complications defined as any complications caused directly or indirectly by the device. Postoperative complication will be classified according to the Clavien-Dindo classification (Grade 1 to Grade 5).

SECONDARY OUTCOMES:
Rate of intraoperative time-out | The day of the procedure
  The rate of intraoperative time-out is defined as a pause in surgical activities lasting at least 2 seconds before clipping and cutting the cystic duct or the cystic artery.
Rate of CVS implementation | The day of the procedure
  The rate of implementation of the CVS will be assessed postoperatively on surgical videos
Surgeons' acceptance | The day of the procedure
  Surgeons' use and acceptance of the technology will be assessed with a specifically designed survey
Patients' acceptance | The day of the procedure
  Patients' acceptability and expectations on the device will be assessed with a specifically designed survey

CONTACTS AND LOCATIONS:
Overall Officials: Silvana PERRETTA, MD, PhD, Principal Investigator — Hopitaux Universitaires de Strasbourg
Locations (1):
- Visceral and Digestive Surgery, Nouvel Hôpital Civil, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No